CLINICAL TRIAL: NCT02415140
Title: Prevalence and Independent Predictors of Depression in COPD
Brief Title: Prevalence and Predictors of Depression in COPD
Status: Completed | Type: Observational
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Tse Hoi Nam, Associate Consultant, Kwong Wah Hospital
Other Study IDs: KW/EX-13-142 (70-02)
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Depression; COPD
MeSH Terms: conditions — Depression; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- COPD: Spirometry confirmed COPD patients
  Interventions: Other: Rate of depression
- Control: normal geriatric patients without lung disease
  Interventions: Other: Rate of depression

INTERVENTIONS:
Other: Rate of depression

SUMMARY:
Depression adversely affects quality of life in COPD patients, associated with higher rate of exacerbations, admissions and mortality. However, local prevalence rate of depression in geriatric COPD patients remains unknown.

Though BODE index is superior to FEV1 in prediction of depression in COPD, it is unclear which domain of BODE correlates best with depression. Furthermore, with multiple confounding factors, it's ambiguous that whether frequent exacerbation is an 'independent' predictor for depression among COPD patients.

The objective of this study is i.) to study the local prevalence rate of depression in geriatric COPD patients, ii.) to identify risk factors for depression especially looking at the any independent relationship between frequent exacerbations, various domains of BODE index and depression.

DETAILED DESCRIPTION:
This study is a multi-centers, cross-sectional study, conducted in Kwong Wah Hospital and Wong Tai Sin Hospital, Hong Kong SAR. Age and comorbidity-matched COPD and control subjects were recruited from clinics. Depressive symptoms were measured by a validated Chinese version of Geriatric Depression Scale short form (GDS - 15 items) with 2 cut-off points. A score of 8 or above was considered significant depressive symptoms while the cut off score of 5 or above was for patients with mild depressive symptoms. Prevalence rates of depressive symptoms were measured in both COPD and control groups. Predictors for depression (GDS = or> 8) were determined using univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above,
* with stable COPD suggested clinically and
* post-bronchodilator spirometry FEV1/FVC ratio <0.7.

Exclusion Criteria:

* Patients were excluded if they had co-existing pulmonary diseases like active pulmonary tuberculosis, interstitial lung diseases etc;
* if they were too demented or physically incapacitated to participate e.g wheelchair-bound for bedbound.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients with spirometry confirmed airflow limitation
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression (Prevalence rate) | 1 year